CLINICAL TRIAL: NCT03903536
Title: Treatment of Thrombosed External Hemorrhoids: Comparison of the Thrombectomy and Local Excision Procedures in Terms of Results and Outcome: A Multi-Centre, International, Prospective Cohort Study
Brief Title: Thrombosed External Hemorrhoids: Comparison of the Thrombectomy and Local Excision Procedures in Terms of Results and Outcome (TEH)
Acronym: TEH
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ali Yalcinkaya, Principal Investigator, Gazi University
Other Study IDs: GaziGenelCerrahiTEH
Record Dates: First submitted 2019-04-01; First posted 2019-04-04 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Thrombosed External Hemorrhoid
MeSH Terms: interventions — Thrombectomy; Hemorrhoidectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Thrombectomy: Patients with thrombosed external hemorrhoids undergoing thrombectomy
  Interventions: Procedure: Thrombectomy
- Local excision/ Hemorrhoidectomy: Patients with thrombosed external hemorrhoids undergoing local excision/ hemorrhoidectomy
  Interventions: Procedure: Hemorrhoidectomy

INTERVENTIONS:
Procedure: Thrombectomy — A small procedure where surgeons make a cut in the hemorrhoid and drain the blood.
  Groups: Thrombectomy
Procedure: Hemorrhoidectomy — A surgery to remove the hemorrhoid, including the blood vessels and clot.
  Groups: Local excision/ Hemorrhoidectomy

SUMMARY:
The primary aim of the current study is to evaluate and compare 6-month complication rates after thrombectomy and local excision treatments.

The investigators aim to compare thrombectomy and local excision treatments in many different aspects:

* The investigators will follow these patients for 6 months by scheduling follow-up visits (or by phone if the patient cannot attend) 4 times during this period (1st week, 1st month, 3rd month, 6th month).
* The investigators will examine bleeding, pain, anal stricture/stenosis, infection, time until return to normal daily activity, relapse and incontinence after treatment
* To assess quality of life outcomes, the investigators use the 36-Item Short Form Health Survey (SF-36). These measures rely upon patient self-reporting and are utilized for routine monitoring and assessment of care outcomes in patients.
* The investigators will use the Wexner incontinence score for assessment of incontinence.

In each hospital, medical students, residents and surgeons can be involved in the study. In the following 6-month period, all collaborators will be collecting the data of the patients who have been operated for external hemorrhoids via the thrombectomy or local excision procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosis with thrombosed external hemorrhoids.
* Providing a written informed consent form for the surgeries and for participation in the study
* Patients aged 18 years and over should be included

Exclusion Criteria:

* Patients younger than 18 years of age,
* Pregnancy
* Patients who have a history of cancer or inflammatory bowel disease(IBD)
* Patients who have a history of anorectal fistula
* Patients with metabolic disorders
* Patients with alcohol or substance addiction
* Patients who refuse to participate in the study and do not provide informed consent
* Patients who, at any stage of the study, indicate that they want to leave the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who apply (or are referred) to general surgery departments and are diagnosis with thrombosed external hemorrhoids will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
6-month complication rate | 6 months from operation
  * The investigators will follow these patients for 6 months by scheduling follow-up visits (or by phone if the patient cannot attend) 4 times during this period (1st week, 1st month, 3rd month, 6th month).
  * The investigators will examine anal bleeding(exist or not), pain(exist or not), anal stricture/stenosis(exist or not, its severity), infection(exist or not), time until return to normal daily activity, relapse and incontinence after treatment.
  * The investigators will use the Wexner incontinence score for assessment of incontinence.
  * The investigators will measure the internal diameter of anal canal for the assessment of anal stenosis and its severity. When the internal diameter of anal canal is less than 0.5 cm, it is severe stenosis and when the diameter is 0.5-1 cm stenosis is moderate and 1-1.5 cm diameter is known as mild stenosis.
6-month quality of life outcomes | 6 months from operation
  Quality of life outcomes within 6 months of surgical procedure. To assess quality of life outcomes, the investigators use the 36-Item Short Form Health Survey (SF-36). The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 - 100. Lower scores = more disability, higher scores = less disability.
  Sections:
  * Vitality
  * Physical functioning
  * Bodily pain
  * General health perceptions
  * Physical role functioning
  * Emotional role functioning
  * Social role functioning
  * Mental health

CONTACTS AND LOCATIONS:
Overall Officials: Sezai Leventoglu, Professor, Study Chair — Gazi University Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Gazi University, Ankara
  - Yildirim Beyazit University Yenimahalle Training and Research Hospital, Ankara

IPD SHARING:
Plan to Share IPD: Yes
Derived anonymised data at the patient-level may be able to be made available for sharing
Supporting Information: Study Protocol, SAP
Time Frame: Following publication of the main results